CLINICAL TRIAL: NCT00001856
Title: Live Donor Renal Donation for Allotransplantation
Brief Title: Live Donors for Kidney Transplants
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990107; 99-DK-0107
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2014-05-30

CONDITIONS: Kidney Transplantation
Keywords: Living Donor; Transplantation; Nephrectomy

SUMMARY:
On a yearly basis there are approximately 12,000 kidney transplants in the United States. Presently there are approximately 40,000 patients awaiting a transplant with only 5,000 available donors. Due to the obvious difference between organ supply and demand, live donors have become a standard source of kidneys for transplantation.

Research has proven that kidneys from living donors are superior to cadaveric donors (kidneys harvested from a deceased individual). Kidneys from living donors are not exposed to extremely low temperature that could increase post-operative problems. They are less likely to experience rejection and there is a decreased likelihood that a patient will have to undergo post-operative dialysis.

The objective of this study is to promote the enrollment of healthy individuals to serve as kidney donors for patients undergoing research kidney transplantation at the NIH. Potential donors will be screened to make sure they are able to survive with a single kidney without significant medical risk. Additional tests will be taken to establish compatibility with the recipient. Compatible donors will be evaluated to determine which kidney is suitable for transplantation. Both the donation and transplantation procedure will be conducted on the same day. Appropriate post-operative care and follow-up will be provided at the Clinical Center.

DETAILED DESCRIPTION:
This protocol is designed to facilitate the enrollment of healthy individuals to serve as renal allograft donors for subjects undergoing protocol renal transplantation at the NIH. Donation will be allowed for altruistic purposes only.

ELIGIBILITY:
* INCLUSION CRITERIA:

Willingness to donate without evidence of secondary gain, coercion, or conflict of interest.

Age greater than or equal to 18 years

ABO compatible with recipient

Normal renal function with a 24hr creatinine clearance greater than 80ml/min/1.73m(2).

Willingness and legal ability to give informed consent

Recipient is enrolled in a NIH protocol for transplantation or has been established as a candidate for receipt of an altruistic or paired donation through the Washington Regional Organ Procurement Agency donor program.

EXCLUSION CRITERIA:

Hypertension

Pregnancy

History of stroke

Active tuberculosis

History of active malignancies except basal cell carcinoma of the skin.

Major anticipated illness or organ failure incompatible with survival after nephrectomy

Functionally significant coronary artery disease.

Active kidney stones

Proteinuria (greater than 250mg/24hr)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 1999-05-17; Study Completion 2014-05-30

CONTACTS AND LOCATIONS:
Overall Officials: Monique E Cho, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cecka JM, Terasaki PI. The UNOS Scientific Renal Transplant Registry. Clin Transpl. 1993:1-18. PMID 7918142
- [Background] Cicciarelli J. Living donor kidney transplants. Clin Transpl. 1988:293-9. PMID 3154482
- [Background] Matas AJ, Gillingham KJ, Sutherland DE. Half-life and risk factors for kidney transplant outcome--importance of death with function. Transplantation. 1993 Apr;55(4):757-61. doi: 10.1097/00007890-199304000-00014. PMID 8475549